CLINICAL TRIAL: NCT01278043
Title: Incidence, Predictors and Impact of Response Variability to Oral Dual Antiplatelet Therapy, as Measured by Point-of-care Platelet Aggregometry, Following Percutaneous Coronary Intervention
Brief Title: Antiplatelet Response, Interval Variability & Events in Percutaneous Coronary Intervention (ARIVE-PCI) Registry
Acronym: ARIVE-PCI
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-222-A
Record Dates: First submitted 2011-01-10; First posted 2011-01-17 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
Keywords: Antiplatelet; Percutaneous Coronary Intervention; Coronary artery disease; Antiplatelet Response, Interval Variability & Events in Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects in this study have recently had or are scheduled for a percutaneous coronary intervention (PCI) as part of their normal, routine medical care. This procedure should restore the blood flow in the vessels of the heart.

One complication that can occur after a PCI procedure is blood clotting and narrowing of the artery in the area that was treated. This can result in a decrease in the blood flow to the heart. To avoid this complication, patients are given antiplatelet or "blood-thinning" drugs such as aspirin and clopidogrel as part of their routine care after this procedure.

For this research study, the investigators would like to take blood samples from subjects at 3 different time points while they are taking these antiplatelet drugs. The investigators will study the subjects' blood and medical history to help us further our understanding of how these drugs respond in individuals and in certain patient populations. Everyone responds a little differently to medications due to many reasons including our genetic make-up. Genes are passed down from our parents and determine our physical appearance such as the color of our hair and eyes. Differences in our genes may also help explain why some drugs work in some people, but not in others. By studying subjects' blood, medical history, genetic make-up and by recording how the subjects' blood responds over the course of their treatment, the investigators hope to learn more about how our bodies respond when taking these drugs. Additionally, the investigators hope to find better ways to predict who will respond more effectively to these drugs and better ways to monitor how these drugs are working in patients' bodies over time after PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for study participation will be obtained following performance of clinically-indicated PCI
* 18 years old and up
* Subjects must have received an oral load of clopidogrel (600 mg total) and aspirin (325 mg if aspirin naïve or minimum 81 mg if on therapy for ≥ 5 days) over the 24 hours preceding enrollment in order to be eligible.

Exclusion Criteria:

* Patients who are unable or unwilling to provide written informed consent or an accurate medical history,
* patients unwilling to participate in follow-up,
* incarcerated or pregnant patients and patients under 18 years of age will be excluded.
* Additionally patients within 24 hours of discontinuation of eptifibatide or tirofiban infusion or within 2 weeks of abciximab infusion,
* patients on antiplatelet monotherapy and patients currently on cilostazol or dipyridomole will be excluded as will those likely to discontinue dual antiplatelet therapy during the 6-month follow up.
* Patients with active bleeding or recent cerebrovascular accident (CVA, "stroke") (≤1 month) at the time of PCI will be excluded, however patients with a history of CVA, bleeding, anemia or thrombocytopenia are eligible providing the clinically-determined careplan includes long-term dual antiplatelet therapy (DAPT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients undergoing PCI at a single medical center will be enrolled in this prospective, open cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is occurrence of significant interval thienopyridine response variability and/or inhibition of platelet aggregation (IPA)) measured at study entry vs. 1 week vs. 1 month following oral thienopyridine load. | 1 month
The co-primary endpoint is occurrence of absolute thienopyridine hyporesponse at any of the specified timepoints. | 2 years

SECONDARY OUTCOMES:
The secondary endpoint of the study explores the relationship between CYP 2C19 genotypes (ultra-rapid and extensive metabolizers vs. intermediate and poor metabolizers) and thienopyridine response / response variability. | 2 years
Exploratory analyses will assess correlation between point-of-care platelet aggregometry (VerifyNow) and laboratory-based assessment of platelet function via Light Transmittance Aggregometry (LTA). | 2 years
Additional analysis will explore the correlation between antiplatelet response to aspirin (ASA) and thienopyridines with incident major adverse cardiac events (MACE) and bleeding events during a 6 month follow-up period. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Nathan, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States